CLINICAL TRIAL: NCT05827042
Title: Endovascular Thrombectomy Alone Versus Intravenous Thrombolysis Plus Endovascular Thrombectomy on Acute Basilar Artery Occlusion - a Multicenter, Randomized Controlled, Clinical Trial
Brief Title: Endovascular Thrombectomy Alone Versus Intravenous Thrombolysis Plus Thrombectomy on Acute Basilar Artery Occlusion
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATTENTION IV
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Basilar Artery Occlusion; Acute Cerebrovascular Accident; Stroke Due to Basilar Artery Occlusion
Keywords: Thrombectomy; thrombolysis
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endovascular thrombectomy alone (Experimental): Patients will receive endovascular thrombectomy without intravenous thrombolysis.
  Interventions: Procedure: Endovascular thrombectomy
- Intravenous thrombolysis plus endovascular thrombectomy (Active Comparator): Patients will receive intravenous alteplase (0.9mg/kg, maximum 90mg) or tenecteplase (0.25mg/kg, maximum 25mg) before endovascular thrombectomy.
  Interventions: Drug: Intravenous thrombolysis; Procedure: Endovascular thrombectomy

INTERVENTIONS:
Drug: Intravenous thrombolysis — Patients will receive intravenous alteplase (0.9mg/kg, maximum 90mg) or tenecteplase (0.25mg/kg, maximum 25mg) before endovascular thrombectomy.
  Other Names: Alteplase or Tenecteplase
  Arms: Intravenous thrombolysis plus endovascular thrombectomy
Procedure: Endovascular thrombectomy — Endovascular thrombectomy

SUMMARY:
To assess the effect of endovascular thrombectomy alone compared to intravenous thrombolysis plus endovascular thrombectomy in acute basilar artery occlusion patients within 4.5 hours from onset on efficacy and safety outcomes.

DETAILED DESCRIPTION:
Two recent randomized, controlled trials from China-ATTENTION (Trial of Endovascular Treatment of Acute Basilar-Artery Occlusion) and BAOCHE (Trial of Thrombectomy 6 to 24 Hours after Stroke Due to Basilar-Artery Occlusion) have shown a significantly beneficial effect of endovascular thrombectomy in patients with an acute symptomatic basilar artery occlusion. The DEVT (Direct Endovascular Treatment versus Standard Bridging Therapy for Acute Stroke Patients with Large Vessel Occlusion in The Anterior Circulation) and DIRECT-MT (Direct Intraarterial Thrombectomy in Order to Revascularize Acute Ischemic Stroke Patients with Large Vessel Occlusion Efficiently in Chinese Tertiary Hospitals Trial) trials showed that endovascular thrombectomy alone is not inferior to intravenous alteplase bridging with endovascular treatment in terms of achieving 90-day functional independence for stroke patients with large vessel occlusion. However, it is unclear whether endovascular thrombectomy alone is noninferior to intravenous thrombolysis bridging with endovascular thrombectomy for achieving functional independence at 90 days among patients with acute basilar artery occlusion. Therefore, additional studies are needed to explore the potential benefit of endovascular thrombectomy alone in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with posterior circulation ischemic stroke symptoms due to basilar artery occlusion or vertebral artery occlusions that prevent antegrade flow into the basilar artery;
2. Time from stroke onset to randomization within 4.5 hours of estimated time of basilar artery occlusion;
3. Patient's age ≥ 18 years;
4. Presence of basilar artery or vertebral artery occlusion, confirmed by CT Angiography (CTA), MR Angiography (MRA) or Digital Subtraction Angiography (DSA). In case of vertebral artery occlusion, the occlusion must completely prevent antegrade flow into the basilar artery;
5. Patients presenting with acute ischemic stroke eligible to receive both endovascular thrombectomy and intravenous thrombolysis using standard criteria;
6. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥ 10;
7. The patient or patient's legal representative signs the informed consent form.

Exclusion Criteria:

1. CT or MR evidence of intracerebral hemorrhage (the presence of < 10 microbleeds is allowed);
2. Pre-stroke modified Rankin scale (mRS) score ≥ 2;
3. Posterior circulation Acute Stroke Prognosis Early CT Score (PC-ASPECTS) on CT/ CTA-Source Images<6; PC-ASPECTS on magnetic resonance imaging-diffusion weighted imaging (MRI-DWI) <5;
4. Pregnant or lactating women;
5. Allergy to contrast agent or nitinol alloy;
6. Life expectancy<1 year;
7. CTA/MRA/DSA show vascular tortuosity, anatomical variation or artery dissection, which would make it difficult to perform endovascular treatment;
8. Participating in other clinical trials;
9. Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, which can not be controlled by antihypertensive drugs;
10. Genetic or acquired hemorrhagic diathesis, lack of anticoagulant factor; oral anticoagulant with international normalized ratio (INR) > 1.7; or novel oral anticoagulant within prior 48 hours;
11. Blood glucose <50 mg/dl (2.8 mmol/L) or >400 mg/dl (22.2 mmol/L), platelet< 100*109/L;
12. Renal insufficiency defined as serum creatinine >2.0 mg/dl (or 176.8 μ mol/l), glomerular filtration rate <30 mL/min, need for hemodialysis or peritoneal dialysis;
13. Patients who cannot complete 90-day follow-up (such as patients without fixed residence, overseas patients, etc);
14. The patient has acute ischemic cerebral infarction within 3 months from randomization;
15. The patient had a history of or clinical suspicion for cerebral vasculitis or infectious endocarditis;
16. The patient has nervous system disease or mental disorder before stroke onset, which may affect the assessment of their condition;
17. CT or MR examination showed large cerebellar infarction with obvious space occupying effect and compression of the fourth ventricle;
18. Patients with extensive bilateral thalamic or extensive bilateral brainstem infarction on CT or MR examination;
19. CTA/MRA/DSA show both anterior and posterior circulation large vessel occlusion;
20. Patients with intracranial tumors (except small meningiomas);
21. Patients who received intravenous thrombolytics treatment before the randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-2 at day 90 (±14 days) | 90 (± 14 days) after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0-3 at day 90 (±14 days) | 90 (± 14 days) after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Proportion of patients with modified Rankin Score 0-1 at day 90 (±14 days) | 90 (± 14 days) after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Proportion of patients with modified Rankin Score 0-4 at day 90 (±14 days) | 90 (± 14 days) after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Ordinal Shift analysis of modified Rankin Score at day 90 (±14 days) | 90 (± 14 days) after procedure
  The modified Rankin Score is an ordinal hierarchical scale ranging from 0 to 6, with higher scores indicating more severe disability.
Score on the National Institute of Health Stroke Scale (NIHSS) at 24 hours | 24 hours after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Score on the NIHSS at 5-7 days or discharge | 5-7 days or discharge after procedure
  The NIHSS is an ordinal hierarchical scale to evaluate the severity of stroke by assessing a patient's performance. Scores range from 0 to 42, with higher scores indicating a more severe deficit.
Score on the EuroQoL 5-dimensions 5-level (EQ5D-5L) at 90 days (±14 days) | 90 (± 14 days) after procedure
  The EQ-5D-5L is a questionnaire designed to assess five dimensions of life quality related to mobility, self-care, usual activities, pain or discomfort, and anxiety or depression (range: 0.39 to 1, with a higher score indicating a higher quality of living)
level of activities of daily living (Barthel index, BI) at 90 days (±14 days) | 90 (± 14 days) after procedure
  The Barthel Index is an ordinal scale for measuring performance of patients'self-care activities of daily living. Scores range from 0 to 100, with 0 indicating severe disability and 95 or 100 indicating no disability that interferes with daily activities.
Successful reperfusion (Extended thrombolysis in cerebral infarction [eTICI] score 2b50-3) on digital substraction angiography (DSA) prior to thrombectomy | within 5 minutes at angiography
  Evaluate effect of intravenous thrombolysis on reperfusion
Successful reperfusion on final angiography of thrombectomy | Within 5 minutes at final angiography of thrombectomy
  Evaluate effect of thrombectomy on reperfusion
Successful recanalization on CT or MR angiography within 72 hours | Within 72 hours after procedure
  Evaluate vascular patency after treatment
Infarct volume (Posterior Circulation Acute Stroke Prognosis Early Computed Tomography Score, PC-ASPECTS) evaluated on CT or MRI within 72 hours | Within 72 hours after procedure
  PC-ASPECTS=10 indicates a normal scan, PC-ASPECTS=0 indicates early ischemic changes or hypoattenuation in all above territories. 1 or 2 points each are subtracted for early ischemic changes or hypoattenuation in: left or right thalamus, cerebellum or posterior cerebral artery territory, respectively (1 point); any part of midbrain or pons (2 points)

OTHER OUTCOMES:
Symptomatic intracerebral hemorrhage (sICH) within 72 hours | Within 72 hours after procedure
  Symptomatic intracranial hemorrhage defined as local or remote parenchymal hemorrhage type 2, subarachnoid hemorrhage, or intraventricular hemorrhage that led to death or was observed on an imaging scan obtained 24 to 72 hours after treatment, combined with a neurologic worsening of at least 4 points from baseline on the NIHSS or from the lowest NIHSS score between baseline and 24 hours, or death from any cause within 90 days.
Any intracerebral hemorrhage within 72 hours | Within 72 hours after procedure
  Evaluate intracerebral hemorrhage
Overall mortality at 7 (± 2 days) and 90 (± 14 days) | 7 (± 2 days) and 90 (± 14 days) after procedure
  Evaluate death rate

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, MD, Study Chair — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China